CLINICAL TRIAL: NCT03943446
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase 2a Study to Evaluate the Safety, Tolerability, and Early Proof of Concept of TAK-018 for the Prevention of Postoperative Crohn's Disease Recurrence
Brief Title: A Study of TAK-018 in Preventing the Recurrence of Crohn's Disease After Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to discontinue study due to inability to recruit the expected number of subjects within the requisite time period.
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TAK-018-2001; 2019-000886-19 (EudraCT Number); U1111-1225-5064 (Registry Identifier: WHO); NR266345 (Registry Identifier: IRAS); NL71098.018.19 (Registry Identifier: CCMO)
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Results first posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Crohn Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): TAK-018 placebo-matching tablets, orally, twice daily (BID) for up to 27.7 weeks.
  Interventions: Drug: TAK-018 Placebo
- TAK-018 0.30 g Low Dose (Experimental): TAK-018 0.30 gram (g), tablets, orally, BID for up to 31.7 weeks.
  Interventions: Drug: TAK-018
- TAK-018 1.5 g High Dose (Experimental): TAK-018 1.5 g, tablets, orally, BID for up to 26.1 weeks.
  Interventions: Drug: TAK-018

INTERVENTIONS:
Drug: TAK-018 — TAK-018 immediate-release tablets.
  Other Names: Sibofimloc
  Arms: TAK-018 0.30 g Low Dose; TAK-018 1.5 g High Dose
Drug: TAK-018 Placebo — TAK-018 placebo-matching tablets.
  Arms: Placebo

SUMMARY:
The main aim is to see if TAK-018 reduces the recurrence of intestinal inflammation after abdominal resection surgery in adults with Crohn's disease.

Participants will take either TAK-018 or placebo tablets by mouth, 2 times each day for up to 26 weeks after surgery. The placebo looks like TAK-018 but will not have any medicine in it.

Participants will have 6 study visits while receiving treatment. Visits 1 and 6 will be conducted at the study clinic. The others can be in the clinic or at the participant's home. Follow-up will occur 4 weeks after final treatment.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-018 (Sibofimloc). TAK-018 is used for the prevention of postoperative CD recurrence. This study will evaluate the efficacy of TAK-018 in reducing endoscopic recurrence of intestinal inflammation in postoperative participants with CD after planned laparoscopic ileocecal resection with primary anastomosis.

The study will enroll approximately 96 participants. Participants will be randomly assigned (by chance, like flipping a coin) in 1:1:1 ratio to one of the three treatment groups-which will remain undisclosed to the participants and study doctor during the study (unless there is an urgent medical need):

* TAK-018 0.30 g Low dose
* TAK-018 1.5 g High dose
* Placebo

All participants will be asked to take the tablets twice daily immediately after a meal (that is, breakfast and dinner) with water, approximately 8 to 12 hours apart.

Participants will have flexibility to either to opt for home health care (HHC) solutions at Screening, Week 3, Week 6, Week 12, Week 18 and Week 30 or travel to the clinic for all scheduled visits per protocol as permitted by local regulations. This flexible approach is designed in response to health care delivery challenges presented by the coronavirus disease (COVID-19) pandemic and to provide additional flexibility during the course of the trial. Assessments after surgery and endoscopy at Week 26 will be conducted at the clinic. All other study visits may be conducted by telehealth and home health care (HHC).

This multi-center trial will be conducted in the United States, United Kingdom, France, Austria and Germany. The overall time to participate in this study is approximately 34 weeks. Participants will make final visit to the clinic or can opt for HHC visit at Week 30 (30 days after the Week 26 endoscopy) for safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Must have a documented diagnosis of CD confirmed by endoscopic biopsy before resection or by tissue obtained at resection.
2. Planned to undergo a laparoscopic ileocecal resection with primary anastomosis within 72 hours before randomization Day 1. Confirmation that no active disease has been left behind after resection will be based on surgeon's documentation in the operative report.
3. With postoperative discontinuation of all concomitant medications specifically related to the treatment of CD. This includes anti-tumor necrosis factor-alpha (TNF-α) and anti-integrin therapy, anti- interleukin (IL) 12/23, thiopurines and other immunomodulators, steroids, 5-minosalicylates, and prophylactic use of antibiotics for the prevention of postoperative recurrence such as metronidazole.
4. Has resumed oral intake and is capable of swallowing tablets within 72 hours after surgery.

Exclusion Criteria:

1. Has active perianal CD.
2. Has had >3 previous surgical procedures for CD.
3. Has macroscopically active CD that was not resected at the time of surgery as documented in the surgeon's operative report.
4. With small bowel resection that exceeds 100 centimeter (cm) or a participant who is considered at risk of short bowel syndrome by the surgeon or investigator.
5. Has active or latent tuberculosis, regardless of treatment history, as evidenced by any of the following: history of tuberculosis, OR positive QuantiFERON test or 2 successive indeterminate QuantiFERON tests, OR a tuberculin skin test reaction ≥10 millimeter (mm) (≥5 mm in participants receiving the equivalent of >15 milligram per day (mg/day) prednisone).
6. Has chronic hepatitis B (hepatitis B surface antigen positive, or positive for both hepatitis B surface antibody and hepatitis B core antibody but negative for hepatitis B surface antigen) or hepatitis C infection (evident by viral replication by polymerase chain reaction) within 30 days of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (41):
- United States (23):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Los Angeles, California
  - University of Colorado Hospital Anschutz Cancer Pavilion, Aurora, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - University of Miami Leonard M. Miller School of Medicine, Miami, Florida
  - University of South Florida/USF Health, Tampa, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - NYU Langone Inflammatory Bowel Disease Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Atrium Health, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt Inflammatory Bowel Disease Clinic, Nashville, Tennessee
  - Houston Methodist Hospital, Houston, Texas
- Austria (2):
  - Medizinische Universitat Innsbruck, Innsbruck, Tyrol
  - Allgemeines Krankenhaus Wien, Vienna, Vienna
- France (6):
  - Les Hopitaux Universitaires de Strasbourg - Hopital Hautepierre, Strasbourg, Alsace
  - Centre Hospitalier Universitaire Estaing, Clermont-Ferrand, Auvergne
  - Hopital Pontchaillou, Rennes, Brittany Region
  - Hopital Saint-Louis, Paris, Il-de-France
  - Hopital Rangueil, Toulouse, Midi-pyrenees
  - Centre Hospitalier Universitaire de Nice Hopital l'Archet, Nice, Provence-Alpes-Côte d'Azur Region
- Germany (6):
  - Universitatsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitatsmedizin Mannheim, Mannheim, Baden-Wurttemberg
  - Klinikum Luneburg, Lüneburg, Lower Saxony
  - Evangelisches Krankenhaus Kalk, Cologne, North Rhine-Westphalia
  - Klinikum Sankt Georg GmbH, Leipzig, Saxony
  - Krankenhaus Waldfriede, Berlin
- United Kingdom (4):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, England
  - London North West Healthcare NHS Trust, Harrow, England
  - Saint Helens and Knowsley Teaching Hospitals NHS Trust, Prescot, England
  - NHS Greater Glasgow and Clyde, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f6b603b4db2bf003ab4a2e7

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 18 investigative sites in the United States, Australia, Germany, France and United Kingdom from 4 August 2020 to 25 August 2022.
Pre-assignment Details: Participants with Crohn's disease (CD) who had undergone a planned laparoscopic ileocecal resection received TAK-018 for prevention of the recurrence of postoperative CD. The participants were randomized in 1:1:1 ratio to three treatment groups i.e. TAK-018 low dose, TAK-018 high dose, or placebo for a 26-week treatment period.
Groups:
- TAK-018 0.30 g Low Dose: TAK-018 0.30 g, tablets, orally, BID for up to 31.7 weeks.
Period: Overall Study
Arm/Group | Placebo | TAK-018 0.30 g Low Dose | TAK-018 1.5 g High Dose
Started | 12 | 11 | 11
Pharmacokinetic (PK) Analysis Set (PK analysis set included participants from the safety analysis set with at least 1 reported PK concentration.) | 12 | 11 | 11
Completed | 5 | 7 | 4
Not Completed | 7 | 4 | 7
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Study Terminated by Sponsor | 1 | 2 | 1
Not completed — Reason not Specified | 5 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants to whom study treatment had been assigned by randomization and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TAK-018 0.30 g Low Dose | TAK-018 1.5 g High Dose | Total
Number analyzed (Participants) | 12 | 11 | 11 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.97 (13.133) | 37.42 (16.179) | 39.25 (11.297) | 39.97 (13.457)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 3 | 17
  Male | 7 | 2 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 9 | 7 | 10 | 26
  Unknown or Not Reported | 2 | 3 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 7 | 10 | 27
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 1 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 3 | 10
  Austria | 4 | 2 | 2 | 8
  Germany | 1 | 1 | 4 | 6
  United Kingdom | 0 | 0 | 1 | 1
  France | 3 | 5 | 1 | 9
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 171.87 (7.709) | 167.95 (7.692) | 172.57 (8.594) | 170.83 (8.019)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 72.44 (13.514) | 67.61 (15.111) | 77.95 (19.971) | 72.66 (16.394)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per meters squared (kg/m^2)] — BMI was calculated based on the height and weight, using the formula: BMI (kg/m^2) = Weight (kg) / [Height (cm)* 0.01]^2.
  kilogram per meters squared (kg/m^2) | 24.57 (4.617) | 23.92 (5.037) | 26.09 (6.175) | 24.85 (5.214)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Endoscopic Recurrence of CD as Assessed by Rutgeerts Grading Scale at Week 26
Description: Endoscopic recurrence (ER) is defined as a Rutgeerts' score ≥ i2. The Rutgeerts scoring is a 5-point scale used to assess endoscopic recurrence at the ileocolonic anastomosis and preanastomotic ileum. The total score ranges from i0 to i4; where i0 = no lesions, i1= ≤ 5 aphthous ulcers, i2= > 5 aphthous ulcers with normal mucosa between lesions or lesions are confined to the anastomosis, i3= diffuse aphthous ileitis with diffusely inflamed mucosa and i4= diffuse inflammation with larger ulcers, nodules, and/or narrowing. Higher score indicates worsening. Percentages are rounded off to the nearest single decimal.
Time Frame: At Week 26
Population: FAS included all participants to whom study treatment had been assigned by randomization and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-018 0.30 g Low Dose | TAK-018 1.5 g High Dose
Number analyzed (Participants) | 12 | 11 | 11
percentage of participants | 91.7 | 81.8 | 90.9
Statistical Analysis 1: Comparison: Placebo vs TAK-018 0.30 g Low Dose; Test type: Superiority; p = 0.590, Fisher Exact; Estimated Difference in ER Rate = -0.10, 95% CI 2-sided [-0.44 to 0.23]
Statistical Analysis 2: Comparison: Placebo vs TAK-018 1.5 g High Dose; Test type: Superiority; p = 1.000, Fisher Exact; Estimated difference in ERR = -0.01, 95% CI 2-sided [-0.34 to 0.31]

2. Secondary Outcome: Percentage of Participants With Fecal Calprotectin (FCP) >135 Microgram Per Gram (mcg/g) at Weeks 3, 6, 12, 18, 26 and 30
Description: Stool samples were collected for analysis of fecal calprotectin, a biomarker of intestinal inflammatory activity. Percentages are rounded off to the nearest single decimal.
Time Frame: At Weeks 3, 6, 12, 18, 26 and 30
Population: FAS included all participants to whom study treatment had been assigned by randomization and received at least 1 dose of study drug. Overall number of participants analyzed is the number of participants available for analyses. Number analyzed indicates number of participants available for analysis at the given timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-018 0.30 g Low Dose | TAK-018 1.5 g High Dose
Number analyzed (Participants) | 11 | 8 | 7
percentage of participants
  At Week 3: number analyzed (Participants) | 9 | 8 | 7
  At Week 3 | 55.6 | 75.0 | 42.9
  At Week 6: number analyzed (Participants) | 11 | 8 | 6
  At Week 6 | 27.3 | 50.0 | 83.3
  At Week 12: number analyzed (Participants) | 9 | 8 | 6
  At Week 12 | 44.4 | 37.5 | 33.3
  At Week 18: number analyzed (Participants) | 8 | 6 | 5
  At Week 18 | 75.0 | 50.0 | 60.0
  At Week 26: number analyzed (Participants) | 7 | 4 | 4
  At Week 26 | 71.4 | 75.0 | 50.0
  At Week 30: number analyzed (Participants) | 5 | 6 | 4
  At Week 30 | 40.0 | 66.7 | 25.0

3. Secondary Outcome: Ctrough: Observed Plasma Trough Concentrations of TAK-018
Time Frame: Pre-dose and at multiple time points (up to 12 hours) post-dose at Week 3
Population: Pharmacokinetic (PK) analysis set included participants from the safety analysis set with at least 1 reported PK concentration. Overall number of participants analyzed is the number of participants available for analyses.
Measure: Mean (Standard Deviation); unit: milligrams per Litre (mg/L)
Arm/Group | TAK-018 0.30 g Low Dose | TAK-018 1.5 g High Dose
Number analyzed (Participants) | 9 | 5
milligrams per Litre (mg/L) | 13.8 (9.39) | 36.2 (21.7)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 30 days following last dose of study drug (up to 35.98 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Placebo: TAK-018 placebo-matching tablets, orally, BID for up to 27.7 weeks.
Arm/Group | Placebo | TAK-018 0.30 g Low Dose | TAK-018 1.5 g High Dose
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/12 | 4/11 | 2/11
Other Adverse Events (participants affected / at risk) | 11/12 | 6/11 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | TAK-018 0.30 g Low Dose (N=11) | TAK-018 1.5 g High Dose (N=11)
Abdominal abscess (Infections and infestations) | 1 | 0 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Inflammation (General disorders) | 0 | 1 | 0
Mesenteric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | TAK-018 0.30 g Low Dose (N=11) | TAK-018 1.5 g High Dose (N=11)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 1
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 0 | 1
C-reactive protein increased (Investigations) | 3 | 2 | 1
COVID-19 (Infections and infestations) | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0
Faecal calprotectin increased (Investigations) | 3 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 1 | 3
Neuralgia (Nervous system disorders) | 0 | 0 | 1
Peripheral swelling (General disorders) | 1 | 0 | 0
Platelet count increased (Investigations) | 1 | 1 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Red blood cell count decreased (Investigations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Tinea versicolour (Infections and infestations) | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0 | 2

LIMITATIONS AND CAVEATS:
This study is terminated as the sponsor decided to discontinue study due to inability to recruit the expected number of participants within the requisite time period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/46/NCT03943446/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/46/NCT03943446/SAP_001.pdf